CLINICAL TRIAL: NCT00004422
Title: Intravenous Pertussis Immune Globulin in Patients With Severe Childhood Pertussis Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13322; IWK-FDR001044; P9701
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-06

CONDITIONS: Pertussis; Whooping Cough
Keywords: bacterial infection; immunologic disorders and infectious disorders; pertussis; rare disease
MeSH Terms: conditions — Whooping Cough; Bacterial Infections; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immune globulin

SUMMARY:
OBJECTIVES:

Assess the efficacy of a single infusion of a high titer pertussis immune globulin for the treatment of severe pertussis in children.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are randomized to receive an infusion of either pertussis immune globulin or placebo (0.9% saline).

Patients are followed every 2 weeks for up to 6 months.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
* Documented infection with Bordetella pertussis

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174
Dates: Start 1997-08; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Halperin, Study Chair — IWK Health Centre